CLINICAL TRIAL: NCT07245381
Title: A Pilot Study to Investigate the Use of Alendronate to Reduce the Risk of Pelvic Insufficiency Fractures in Cervical Cancer Patients Treated With Chemotherapy and Radiation Therapy
Brief Title: Alendronate to Reduce Pelvic Insufficiency Fractures in Cervical Cancer Patients Undergoing Chemoradiation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Itay GoorAryeh (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Itay GoorAryeh, Head of the Pain Clinic, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1509-24-SMC
Record Dates: First submitted 2025-07-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Cervix Cancer
Keywords: Chemo-Radiotherapy; Alendronate; Cancer of the Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Cancer of the Cervix Treated with Chemo-Radiotherapy (Experimental): Age: Patients must be 18 years of age or older.
  * Diagnosis:Patients diagnosed with non-metastatic cervical cancer stages IB2 to IVA, as per the FIGO staging system.
  * Treatment Plan: Patients scheduled to undergo definitive chemo-radiotherapy or adjuvant chemo-radiotherapy post-surgery.
  * Bone Health: No history of osteoporosis or previous treatment with bisphosphonates or other bone-modifying agents.
  * Pain Assessment: Patients experiencing bone pain or at risk of developing pelvic insufficiency fractures, despite current standard of care.
  * Recent Imaging: Patients must have undergone recent imaging (CT, PET, or MRI) within the last 3 months to confirm the absence of bone metastases.
  * Compliance: Patients must be able to comply with the study protocol and follow-up schedule. Psychological, familial, sociological, or geographical conditions that could hamper compliance need to be evaluated and discussed before trial registration.
  * Consent: Patients must provide written informed co
  Interventions: Drug: Alendronate 70mg weekly

INTERVENTIONS:
Drug: Alendronate 70mg weekly — the Use of Alendronate to Reduce the Risk of Developing Pelvic Insufficiency Fractures in Patients with Cancer of the Cervix Treated with Chemo-Radiotherapy

SUMMARY:
Primary Objective

- Proof of concept: To evaluate the efficacy of alendronate in preventing pelvic insufficiency fractures (PIFs) in cervical cancer patients treated with chemo-radiotherapy over the short and long term. This objective will assess both the immediate and sustained effects of the drug on bone integrity through periodic bone mineral density measurements and clinical assessment of fracture incidence.

Secondary Objectives

* To assess the safety and tolerability of alendronate: This will involve monitoring and documenting any acute and chronic side effects associated with alendronate use in this patient population, including but not limited to gastrointestinal issues, renal function impairment, and osteonecrosis of the jaw.
* To document and analyze changes in quality of life: Using validated quality of life instruments, this objective will track changes in patient-reported outcomes, focusing on aspects such as pain levels, physical function, and overall well-being. This will help determine if the intervention not only prevents fractures but also contributes positively to the patients' quality of life during and after treatment.
* To explore correlations between patient-specific factors and treatment efficacy: This objective aims to understand how variables such as age, cancer stage, previous treatment history, and baseline bone health might influence the effectiveness of alendronate in preventing PIFs and enhancing bone mineral density.

DETAILED DESCRIPTION:
Primary Objective

- Proof of concept: To evaluate the efficacy of alendronate in preventing pelvic insufficiency fractures (PIFs) in cervical cancer patients treated with chemo-radiotherapy over the short and long term. This objective will assess both the immediate and sustained effects of the drug on bone integrity through periodic bone mineral density measurements and clinical assessment of fracture incidence.

Secondary Objectives

* To assess the safety and tolerability of alendronate: This will involve monitoring and documenting any acute and chronic side effects associated with alendronate use in this patient population, including but not limited to gastrointestinal issues, renal function impairment, and osteonecrosis of the jaw.
* To document and analyze changes in quality of life: Using validated quality of life instruments, this objective will track changes in patient-reported outcomes, focusing on aspects such as pain levels, physical function, and overall well-being. This will help determine if the intervention not only prevents fractures but also contributes positively to the patients' quality of life during and after treatment.
* To explore correlations between patient-specific factors and treatment efficacy: This objective aims to understand how variables such as age, cancer stage, previous treatment history, and baseline bone health might influence the effectiveness of alendronate in preventing PIFs and enhancing bone mineral density.

ELIGIBILITY:
Inclusion Criteria:Age: Patients must be 18 years of age or older.

* Diagnosis:Patients diagnosed with non-metastatic cervical cancer stages IB2 to IVA, as per the FIGO staging system.
* Treatment Plan: Patients scheduled to undergo definitive chemo-radiotherapy or adjuvant chemo-radiotherapy post-surgery.
* Bone Health: No history of osteoporosis or previous treatment with bisphosphonates or other bone-modifying agents.
* Pain Assessment: Patients experiencing bone pain or at risk of developing pelvic insufficiency fractures, despite current standard of care.
* Recent Imaging: Patients must have undergone recent imaging (CT, PET, or MRI) within the last 3 months to confirm the absence of bone metastases.
* Compliance: Patients must be able to comply with the study protocol and follow-up schedule. Psychological, familial, sociological, or geographical conditions that could hamper compliance need to be evaluated and discussed before trial registration.
* Consent: Patients must provide written informed consent before participating in the study

Exclusion Criteria:Age: Patients under 18 years of age.

* Performance Status: Patients with an ECOG Performance Status of 2, 3 or 4.
* Bone Metastases: Presence of bone metastases.
* Contraindications to Alendronate: Known contraindications to alendronate, such as esophageal disorders, inability to sit or stand upright for at least 30 minutes, severe renal impairment (creatinine clearance <35 mL/min), or hypersensitivity to any component of the product.
* Concurrent Treatments: Patients receiving other concurrent treatment with bisphosphonates, denosumab, or other bone-modifying agents.
* Special Populations: Pregnant or breastfeeding women, prisoners, and patients with major psychiatric illnesses that could interfere with adherence to study requirements.
* Previous Treatment: Patients who have previously received radiotherapy to the pelvic region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain | Pre -treatment, 5,12 and 24 months post-initiation of therapy
  Use of the numeral rating scale for pain
Quality of life | Pre -treatment and 5,12 and 24 months post-initiation of therapy
  Use of QLQ-C30 scale

SECONDARY OUTCOMES:
Bone Mineral Density | Pre-treatment, 1 year and 2 years post-treatment
  DXA Scan
Blood tests for markers of bone turnover | Pre-treatment
  Calcium and vitamin D levels, CTX(serum C terminal telopeptide),P1NP, Albumin-adjusted Calcium levels, Phosphorus, Estradiol and FSH

IPD SHARING:
Plan to Share IPD: No
All data is part of the Institutional database